CLINICAL TRIAL: NCT02313350
Title: Non-inferiority Trial of Intradiscal Discogel® Versus Surgery in Sciatica Resistant to Conservative Treatment
Brief Title: Intradiscal Discogel® in Resistant Sciatica
Acronym: EDIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: faisability
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gelscom SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: : P130913
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Herniated Disc; Sciatica; Persistent Pain, Leg
Keywords: Sciatica,; herniated disc,; chemonucleolysis.
MeSH Terms: conditions — Intervertebral Disc Displacement; Sciatica | interventions — Intervertebral Disc Chemolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemonucleolysis with Discogel (Experimental): Discogel® is a class III medical device (CE0459 mark on 28/09/2007) constituted by a radiopaque jellified ethanol. Discogel® is provided in a kit containing a 2 ml solution for injection with two disposable 1ml syringes. Discogel® chemonucleolysis for herniated disc-related sciatica is performed under local anesthesia. A volume of 0.9 ml of Discogel® is finally slowly injected during 10 to 15 minutes
  Interventions: Device: Chemonucleolysis with Discogel
- Open discectomy (Active Comparator): surgery : The comparator is open surgical discectomy. The procedure will be performed under general anesthesia. It will consist in removing the disc herniation after exposition and examination of the nerve root
  Interventions: Procedure: open discectomy

INTERVENTIONS:
Device: Chemonucleolysis with Discogel — Discogel® is provided in a kit containing a 2 ml solution for injection with two disposable 1ml syringes, each for single use which is stored at room temperature. Discogel® chemonucleolysis for herniated disc-related sciatica is performed under local anesthesia .
  Arms: Chemonucleolysis with Discogel
Procedure: open discectomy — The comparator is open surgical discectomy. The procedure will be performed under general anesthesia. It will consist in removing the disc herniation after exposition and examination of the nerve root.
  Arms: Open discectomy

SUMMARY:
Sciatica due to herniated disc is a major cause of disability in young adults. Surgery is the gold-standard and the only controlled treatment in case of failure of conservative treatment.

Percutaneous chemonucleolysis with Discogel® may be a valuable alternative to surgery.

In addition, Discogel® chemonucleolysis appears as a relatively innocuous technique which may avoid 2% complications after disc surgery and 5% repeated surgery (according to recent trials).

This will be the first randomized trial comparing Discogel® chemonucleolysis versus surgery in patients with sciatica due to lumbar disc herniation and unresponsive to conservative medical treatments (including epidural steroid injections) Our expectation is that Discogel® chemonucleolysis will avoid surgery in 80% of the patients.

DETAILED DESCRIPTION:
Since chymopapain was taken off the market in 2002, no percutaneous treatment has been proven to be a valuable alternative to surgical discectomy in herniated disk-related sciatica. Intradiscal injection of alcohol was a possibly efficient technique but was not used due to its rapid dissipation and nerve toxicity. The gel, by stabilizing the alcohol into the disc, now makes it effective locally and cancels its nerve toxicity. As a preliminary evaluation, we conducted an open trial with strict methodological criteria to test the efficiency of an intradiscal injection using a new product based on jellified ethanol, Discogel®, in the treatment of nerve root pain due to compression by herniated disk. A 30% improvement in pain VAS was obtained in two thirds of the patients. No complication was encountered. These results prompted us to further investigate the effectiveness of Discogel® chemonucleolysis using a randomized design comparing it to surgery which remains the gold-standard treatment for disk-related sciatica resistant to conservative treatment. Our hypothesis is that chemonucleolysis using Discogel® has suitable efficacy and safety profile for large application in the treatment of persistent herniated disc related sciatica and that it is consequently able to reduce the need of surgery, namely open discectomy, in this indication. New minimally invasive approach of herniated disc-related sciatica is crucial, due to high prevalence and medico-economic impact of the disease. Awaited advances are enrichment of management strategies for herniated disc-related sciatica, earlier recovery of patients unresponsive to first line conservative treatment, reduction of the costs and serious adverse events related with surgery and finally reduction of the costs associated with induced sciatica disability.

Study design:

* Open randomized non-inferiority clinical trial
* Discogel® vs surgery, to be organized within four next weeks after randomization
* Eligible patients who decline participation to the trial will be followed in an observational cohort at the same time-frame as the randomized cohort
* Measurement of compliance with the assigned treatment
* Patients randomized who will delay or decline the assigned treatment will not be excluded from the trial
* Visits at 4, 8, 16, 24 and 52 weeks (evaluation of the main and secondary outcomes)
* Result analysis will be conducted in Intention to treat
* Surgery will be allowed in the Discogel® arm starting at the 16 W visit or before in case of intractable pain or complication.

Study procedures:

Enrollment of patients will be done from the consultations of Rheumatology, Radiology, Surgery and Physical and Rehabilitation Medicine Departments of each study center. Indeed, the inclusion visit will not be done by the physician who will perform the chemonucleolysis, or the surgeon in charge of the patient. After randomization, chemonucleolysis or surgery will be scheduled within the four next weeks. Patients undergoing chemonucleolysis will be hospitalized in day hospital of the Rheumatology / Surgery department of each study center. The procedure of chemonucleolysis will be performed in the corresponding Radiology department or in the usual department. Open discectomy will be performed during a conventional hospitalization in the Surgery department of each study center. Duration of the hospital stay will depend on patient's recovery after surgery. A duration of about one week is expected.

The follow-up of patients will be 52 weeks (5 time points). At each time point, main and secondary outcomes will be evaluated. Questionnaires will be filled out by the patient, before the consultation visit. An independent person (nurse, secretary, clinical research technician..) will be available to help the patient to fill his self questionnaire and check for the accuracy of the patient answers. It is important to note no physician involved in the protocol will participate to the patient evaluation. The physician assessor will be blinded for the result of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* L5 or S1 sciatica due to a herniated disc demonstrated at a MRI performed at a maximum of 8 weeks prior to inclusion
* Leg pain intensity superior to 40mm on a visual-analogue scale despite pain medication (patient with pain level of less than 40 mm and under morphinic treatment, morphine should be first replaced by level 2 medication).
* Leg pain predominant over low back pain
* Duration of sciatica of the current symptomatic episode: from 6 weeks to 40 weeks
* Leg pain resistant to conservative treatment including at least two epidural steroid injections and at least one steroid injection under fluoroscopic guidance, during the current symptomatic episode
* With or without sensitive deficit

Exclusion Criteria:

* - Motricity index < 3/5
* Cauda equinal syndrome
* Sequestered disc herniation visible at MRI
* Calcified/ossified disc herniation visible at MRI
* Intervertebral disc height narrowing > 60%
* Previous back surgery or percutaneous disc treatment at the same intervertebral level
* Psychiatric status precluding patient evaluation
* Pregnancy Any known or documented allergy to one of the components of the Discogel®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of the leg pain score on a 100-mm visual analogue scale | 4, 8, 16, 24 and 52 weeks
  The primary endpoint is the AUC of the leg pain score on a 100-mm visual-analogue scale, assessed by the patient in a self questionnaire at 4, 8, 16, 24 and 52 weeks, calculated by the trapezoidal method.The assessor will be blinded for the result of questionnaires

SECONDARY OUTCOMES:
AUC of back pain score on a visual-analogue scale between 0 and 52 weeks | 4, 8, 16, 24 and 52 weeks
  Pain and questionnaires will be fulfilled by the patient alone and the assessor will be blinded.
AUC of global pain score on a visual-analogue scale between 0 and 52 weeks | 4, 8, 16, 24 and 52 weeks
AUC of Quality of life (SF36) between 0 and 52 weeks | 4, 8, 16, 24 and 52 weeks
Functional disability using the Roland disability questionnaire | at 4, 8, 16, 24, 52 weeks
Assessment of sciatica using the Modified Roland Morris disability scale | at 4, 8, 16, 24, 52 weeks
Medication and other treatment consumption during the one-year Follow-up (FU) | at 4, 8, 16, 24, 52 weeks
Cost-effectiveness in both arms (costs, utilities based on -EQ5D™ scores, cost utility analysis) | 52 weeks
Percentage of surgery in the Discogel® chemonucleolysis arm | 52 weeks
  in Discogel® group only
Number of surgical interventions avoided in the Discogel® arm | 52 weeks
  in Discogel® group Only
Number of assigned treatments finally performed (adherence to assigned treatment in both arms) | 52 weeks
Adverse events | 52 weeks
Number of secondary surgical interventions after Discogel® or after first open discectomy | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johann Beaudreuil, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Rheumatology, Lariboisière Hospital, Paris, France